CLINICAL TRIAL: NCT01841684
Title: A Worldwide, Multicenter, Double-Blind, Randomized, Placebo-Controlled, 12-Week Study to Assess the Efficacy and Tolerability of Anacetrapib When Added to Ongoing Lipid-Lowering Therapy in Adult Patients With Homozygous Familial Hypercholesterolemia (HoFH)
Brief Title: Efficacy and Tolerability of Anacetrapib Added to Ongoing Lipid-Lowering Therapy in Adult Participants With Homozygous Familial Hypercholesterolemia (HoFH) (MK-0859-042)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0859-042; 2012-002434-37 (EudraCT Number)
Record Dates: First submitted 2013-04-24; First posted 2013-04-26 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Hyperlipoproteinemia Type II; Homozygous Familial Hypercholesterolemia
Keywords: HoFH
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Homozygous Familial Hypercholesterolemia | interventions — anacetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anacetrapib (Experimental): Participants receive anacetrapib 100 mg orally once daily for 12 weeks.
  Interventions: Drug: Anacetrapib
- Placebo (Placebo Comparator): Participants receive placebo orally once daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anacetrapib — 100 mg tablet orally, once daily for 12 weeks
  Other Names: MK-0859
  Arms: Anacetrapib
Drug: Placebo — Placebo for anacetrapib orally, once daily for 12 weeks
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and effect of anacetrapib on low-density lipoprotein-cholesterol (LDL-C) when added to ongoing lipid-lowering therapy. The primary hypothesis is that treatment with anacetrapib 100 mg for 12 weeks will lower LDL-C to a greater extent than treatment with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HoFH by genotyping
* If female, cannot be of reproductive potential
* Have been stabilized on statin monotherapy or statin therapy coadministered

with other lipid medications for at least 6 weeks

Exclusion Criteria:

* Severe chronic heart failure defined by New York Heart Association

(NYHA) Classes III or IV

* Uncontrolled cardiac arrhythmias, myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary arterial by-pass graft (CABG), unstable angina or stroke within 3 months prior to Visit 1 or has planned procedures scheduled within first 12 weeks of study
* Uncontrolled endocrine or metabolic disease known to influence serum

lipids or lipoproteins

* Active or chronic hepatobiliary or gall bladder disease
* History of ileal bypass, gastric bypass, or other significant condition

associated with malabsorption

* Human immunodeficiency virus (HIV) positive
* Donated blood products or has had phlebotomy of >300 mL within 8 weeks or intends to donate 250_mL of blood products or receive blood products within the projected duration of the study
* Taking medications that are potent inhibitors or inducers of cytochrome P450 3A4 (CYP3A4), including but not limited to cyclosporine, systemic itraconazole or ketoconazole, erythromycin, clarithromycin, or telithromycin, nefazodone, protease inhibitors, carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, St John's wort) or has discontinued treatment <3 weeks prior. Consumption of >1 liter of grapefruit juice per day is also prohibited.
* Currently participating or has participated in a study with an investigational compound or device within 3 months
* Consume more than 2 alcoholic drinks per day
* Receiving treatment with systemic corticosteroids or systemic anabolic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Percent change from Baseline in Low-density Lipoprotein-Cholesterol (LDL-C) using beta-quantification method | Baseline and Week 12
Number of Participants with Alanine Transaminase (ALT) or Aspartate Aminotransferase (AST) Consecutive Elevations ≥3x Upper Limit of Normal (ULN) | 12 weeks
Number of Participants with Creatine Phosphokinase Elevations ≥10xULN with or without Muscle Symptoms | 12 weeks
Number of Participants with Sodium, Chloride, or Bicarbonate Elevations >ULN or Potassium Levels <Lower Limit of Normal (LLN) | 12 weeks
Number of Participants with Pre-specified Adjudicated Cardiovascular Serious Adverse Events or Death from Any Cause | 12 weeks
Number of Participants with Significant Increase in Blood Pressure | 12 weeks

SECONDARY OUTCOMES:
Percent Change from Baseline in High-density Lipoprotein-cholesterol (HDL-C) | Baseline and Week 12
Percent Change from Baseline in Apolipoprotein A-I (apoA-I) | Baseline and Week 12